CLINICAL TRIAL: NCT06086067
Title: Influence of the Phases of the Menstrual Cycle on Glycemic Control Before, During, and After a Aerobic Exercise in Adult Women With Type 1 Diabetes (TAILOR/1a)
Brief Title: Influence of the Phases of the Menstrual Cycle on Glycemic Control When Performing Aerobic Exercise in Women With T1D
Acronym: TAILOR/1a
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); Ministerio de Ciencia e Innovación, Spain (Other Government); European Regional Development Fund (Other); Universitat Politècnica de València (Other)
Responsible Party: Principal Investigator, Rodrigo Martín-San-Agustin, Professor, University of Valencia
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1586990
Record Dates: First submitted 2023-09-21; First posted 2023-10-17 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: aerobic; woman; glucemic
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Two interventions will be carried out in a single group, being two aerobic sessions, one in luteal phase and another in follicular phase. Because we want to observe both phases in the same menstruation cycle, both aerobic training sessions cannot be randomized.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic session in luteal phase (Experimental): The aerobic exercise session will begin with a 3 min resting period (sitting quietly on the cycle ergometer (0 W), followed by a 3 min warm-up at 40 W and a stepwise intensity increase by 20 W / min (to control for day-to-day variations in exercise response) until the 5% of Pmax from IET above PLTP1 is achieved (i.e. moderate steady state walking or low-intensity running or cycling). This target workload will be maintained for 30 min. Active and passive recovery periods of 3 min each will be the same as the incremental test. This session will be held on day 21 of menstruation.
  Interventions: Other: Aerobic session
- Aerobic session in follicular phase (Experimental): The aerobic exercise session will begin with a 3 min resting period (sitting quietly on the cycle ergometer (0 W), followed by a 3 min warm-up at 40 W and a stepwise intensity increase by 20 W / min (to control for day-to-day variations in exercise response) until the 5% of Pmax from IET above PLTP1 is achieved (i.e. moderate steady state walking or low-intensity running or cycling). This target workload will be maintained for 30 min. Active and passive recovery periods of 3 min each will be the same as the incremental test. This session will be held on day 3 of menstruation.
  Interventions: Other: Aerobic session

INTERVENTIONS:
Other: Aerobic session — This session will consist of an aerobic training session performed on a cycle ergometer.

SUMMARY:
This study corresponds to Task 8.1 of the project "Patient-tailored solutions for blood glucose control in type 1 diabetes- TAILOR" (PID2019-107722RB-C21).

It has been observed in different studies in healthy people that the glucose rate of appearance or disappearance during exercise is attenuated with the coincident rise in estrogen and progesterone during the mid-luteal phase of the menstrual cycle versus the early luteal phase.

The investigators hypothesize that in women with type 1 diabetes, glucose behavior when performing aerobic exercise may be different depending on the phase of the menstruation cycle. This analysis is necessary to improve physical exercise recommendations, both educational and technological, in women with type 1 diabetes, as well as improve the performance of artificial pancreas systems for automatic control of glucose levels under exercise in women.

DETAILED DESCRIPTION:
This study will consist of two aerobic exercise sessions, one conducted at the beginning of the late follicular phase, where maximal estrogen concentration coincides with low progesterone levels, and the other session in the middle of the luteal phase, where peak values of estrogen and progesterone are generally observed.

Prior to the exercise sessions, an incremental exercise test will be performed to determine the working power in the cycle ergometer. At the beginning of the test, subjects will be sit quietly on the cycle ergometer for 3 min (0 W) before they will start the warm-up period of 3 min with cycling at a workload of 40 W. Then, the workload will increase by 20 W every minute until volitional exhaustion. Finally, 3 min active recovery at 40 W followed by 3 min passive recovery (0 W) will be conducted on the cycle ergometer. Lactate turn point 1 (LTP1) and maximum power (Pmax) will be determined in order to prescribe the exercise intensity.

The aerobic exercise session will begin with a 3 min resting period (sitting quietly on the cycle ergometer (0 W), followed by a 3 min warm-up at 40 W and a stepwise intensity increase by 20 W / min (to control for day-to-day variations in exercise response) until the 5% of Pmax from IET above PLTP1 is achieved (i.e. moderate steady state walking or low-intensity running or cycling). This target workload will be maintained for 30 min. Active and passive recovery periods of 3 min each will be the same as the incremental test.

To monitor the impact on blood glucose, blood draws will be performed at initial and every 10 minutes for aerobic sessions. A sample size of n=30 will be chosen.

ELIGIBILITY:
Inclusion criteria:

* age between 18-45 years
* T1D with a diabetes duration for more than 2 years
* glycated hemoglobin (HbA1c) < 8.5% (<69 mmol mol-1)
* stable insulin regimen in the past 6 months with less than 20% change in total insulin daily dose
* multiple daily injections
* weekly physical activity of 90 min or more, but no practicing any sport as amateur or professional.

Exclusion Criteria:

-clinical conditions or use of medications (other than insulin) known to affect glycemic control (e.g., oral/parenteral steroids or metformin, among others).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | The evaluated time points for aerobic exercise will be at 20 and 10 minutes before the session, at the beginning of the training and at 10, 20, and 30 minutes during the interval, and at 10 and 20 minutes after finishing the training.
  Blood glucose (mg/dL) will be measured through blood draws and YSI analysis
Mean interstitial glucose | 24 hours pre-intervention and 24 hours post-intervention
  Mean interstitial glucose (mg/dL) will be measured using the FreeStyle3 as a continuous glucose meter during 6 hours, 12 hours, and 24 hours before and after both exercise sessions.
Glycemic variability | 24 hours pre-intervention and 24 hours post-intervention
  Glycemic variability (measured using the Coefficient of Variation-CV) will be measured using the FreeStyle3 as a continuous glucose meter during 6 hours, 12 hours, and 24 hours before and after both exercise sessions.
Time spent at each glucose range | 24 hours pre-intervention and 24 hours post-intervention
  Time spent at each glucose range [euglycemia (70-180 mg/dL) or Time in range (TIR), level 1 or mild hypoglycemia (54-70 mg/dL), level 2 or severe hypoglycemia (<54 mg/dL), level 1 hyperglycemia (180-250 mg/dL) and level 2 hyperglycemia (>250 mg/dL)] will be measured using the FreeStyle3 as a continuous glucose meter during 6 hours, 12 hours, and 24 hours before and after both exercise sessions.

SECONDARY OUTCOMES:
Lactate | pre-intervention and immediately after the intervention
  Lactate concentration (mmol/L) will be performed through blood extractions and measured using the YSI 2500.
Oestrogens | pre-intervention
  estradiol levels (pg/ml) will be measured through blood extractions and subsequent analysis in the laboratory.
Progesterone | pre-intervention
  Progesterone (ng/mL) will be measured through blood extractions and subsequent analysis in the laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Rodrigo Martin-San Agustin, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cuerda-Del Pino A, Laguna Sanz AJ, Diez JL, Rossetti P, Marco Romero C, Ampudia-Blasco FJ, Bondia J, Martin-San Agustin R. Accuracy of FreeStyle Libre 3 During Moderate-Intensity Continuous Aerobic Exercise at Different Phases of the Menstrual Cycle in Females with Type 1 Diabetes. Diabetes Technol Ther. 2025 Sep;27(9):687-695. doi: 10.1089/dia.2024.0558. Epub 2025 Apr 17. PMID 40256792